CLINICAL TRIAL: NCT03177018
Title: Feasibility of DNA Analysis From Isolated Cardiomyocytes in the Molecular Diagnosis of Arrhythmogenic Right Ventricular Cardiomyopathy/Dysplasia
Brief Title: DNA Analysis From Isolated Cardiomyocytes in the Molecular Diagnosis of Arrhythmogenic Right Ventricular Cardiomyopathy/Dysplasia
Acronym: FA2CM-DVDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC31/15/7731
Record Dates: First submitted 2017-06-02; First posted 2017-06-06 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2023-07

CONDITIONS: Arrhythmogenic Right Ventricular Dysplasia; Arrhythmogenic Right Ventricular Cardiomyopathy
MeSH Terms: conditions — Arrhythmogenic Right Ventricular Dysplasia

STUDY DESIGN:
Intervention Model Description: Exploratory, monocentric and prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Cardiomyocytes collection (Experimental): Patients suffering from arrhythmogenic right ventricular cardiomyopathy/dysplasia cardiac and needing endocardial voltage mapping for disease diagnosis and/or prognosis assessment
  Interventions: Diagnostic Test: Cardiomyocytes collection

INTERVENTIONS:
Diagnostic Test: Cardiomyocytes collection — collect intact cardiomyocytes from which high quality DNA extraction will be achieved

SUMMARY:
The main objective of this study is to assess if it is possible, at the end of endocardial voltage mapping, to accurately collect intact cardiomyocytes and to isolate high quality DNA allowing molecular testing of selected genes involved in arrhythmogenic right ventricular cardiomyopathy/dysplasia.

DETAILED DESCRIPTION:
Arrhythmogenic right ventricular cardiomyopathy/dysplasia is associated with mutations in genes encoding proteins from desmosomes and is characterized by a large expression variability. The classical molecular diagnosis from blood cells fails to identify mutations in around 30% of patients. Probes used for endocardial voltage mapping allow to collect some cardiomyocytes which could be used for DNA analysis.

The aim of this project is to investigate if cardiomyocytes can efficiently be collected during endocardial voltage mapping in patients with arrhythmogenic right ventricular cardiomyopathy/dysplasia. Thirty patients suffering from arrhythmogenic right ventricular cardiomyopathy/dysplasia cardiac and needing endocardial voltage mapping for disease diagnosis and/or prognosis assessment will be included. The main outcome will be the percentage of patients in whom mapping will allow to collect intact cardiomyocytes from which high quality DNA extraction will be achieved. Other outcomes include the identification of new mutational mechanisms as somatic mosaicism in selected genes (PKP2, DSCG2 DSP) and the feasibility of epigenetic analysis of these genes.

ELIGIBILITY:
Inclusion Criteria:

* patients needing endocardial voltage mapping in the context of arrhythmogenic right ventricular cardiomyopathy/dysplasia diagnosed using current criteria

Exclusion Criteria:

* Patient under 18 years, pregnant women and patients under legal protection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-09-13 (Actual); Primary Completion 2018-02-23 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
percentage of patients | inclusion
  Percentage of patients undergoing endocardial voltage mapping for arrhythmogenic right ventricular cardiomyopathy/dysplasia in whom at least one intact cardiomyocyte allowing extraction of high quality DNA will be collected.

SECONDARY OUTCOMES:
Mutation percentage | Inclusion
  Percentage of cases in which a mutation of at least one of three selected genes involved in arrhythmogenic right ventricular cardiomyopathy/dysplasia will be identified
DNA results | Inclusion
  Concordance of results of DNA analysis between blood cells and cardiomyocytes
Epigenetic analysis | Inclusion
  Number of cases where epigenetic analysis of the three selected genes PKP2, DSP, DSG2 from cardiomyocyte DNA could be performed and comparison with DNA methylation observed from blood cells DNA.
Cardiomyocytes number Description: | Inclusion
  Number of intact cardiomyocytes collected in each patient
Percentage of cardiomyocytes | Inclusion
  Percentage of cardiomyocytes from which isolation of high quality DNA will be achieved

CONTACTS AND LOCATIONS:
Overall Officials: Philippe MAURY, MD, Principal Investigator — University Hospital, Toulouse
Locations (2):
- France (2):
  - Cardiology-rytmology service, Paris
  - University Hospital Toulouse - Cardiology Department, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Maury P, Ader F, Lhuillier E, Martins F, Beneyto M, Gales C, Villard E, Duboscq-Bidot L, Gandjbakhch E, Guilbeau-Frugier C. Human DNA Extraction and Sequencing From Cardiomyocytes Collected by Catheter-Based Aspiration. J Am Coll Cardiol. 2024 Jul 30;84(5):490-492. doi: 10.1016/j.jacc.2024.05.037. No abstract available. PMID 39048282